CLINICAL TRIAL: NCT01457755
Title: A Long Term Follow-up Registry for Subjects Who Achieve a Sustained Virologic Response to Treatment in Gilead-Sponsored Trials in Subjects With Chronic Hepatitis C Infection
Brief Title: Gilead Sustained Virologic Response (SVR) Registry
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-248-0122; 2011-000945-19 (EudraCT Number)
Record Dates: First submitted 2011-10-04; First posted 2011-10-24 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; HCV; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; Tegobuvir; Registry; HCV RNA; Treatment experienced; Treatment naive; GS 9451; GS 5885; GS 7977; GS 5816; Sofosbuvir; Sovaldi™; SOF; Ledipasvir; LDV
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
This Registry is designed to provide long term clinical and virologic follow up in participants who have achieved sustained virologic response (SVR) while participating in a previous Gilead sponsored hepatitis C virus (HCV) study. This long term follow up study is observational and no treatment is provided for HCV.

ELIGIBILITY:
Key Inclusion Criteria:

* Have previously participated in a Gilead-sponsored hepatitis C study and received at least one Gilead oral antiviral agent (OAV)
* Have achieved SVR in a Gilead-sponsored study, as defined in the original treatment protocol
* Provide written, informed consent
* Be willing and able to comply with the visit schedule and protocol-mandated procedures

Key Exclusion Criteria:

* Individuals planning to start a new course of hepatitis C therapy including any investigational drug or device during the course of the follow-up Registry
* History of clinically significant illness or any other major medical disorder that may interfere with follow up, assessments, or compliance with the protocol

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have achieved sustained virologic response (SVR) while participating in a previous Gilead sponsored HCV study.
Sampling Method: Non-Probability Sample
Enrollment: 6625 (Actual)
Dates: Start 2012-04-13 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Proportion of participants maintaining SVR at Week 144 by treatment regimen | Week 144

SECONDARY OUTCOMES:
Proportion of participants with detectable HCV RNA due to reemergence of preexisting virus through Week 144 by treatment regimen | Up to 144 weeks
Proportion of participants with detectable HCV resistance mutations through Week 144 by treatment regimen | Up to 144 weeks
Proportion of participants with detectable HCV RNA due to reinfection through Week 144 by treatment regimen | Up to 144 weeks
Liver disease progression | Up to 144 weeks
  Liver disease progression is a composite endpoint measured by laboratory parameters (alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, albumin, platelets, prothrombin time (PT) and α-fetoprotein) and observed or reported clinical signs and symptoms.
Proportion of participants who develop hepatocellular carcinoma (HCC) through Week 144 by treatment regimen | Up to 144 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (318):
- United States (161):
  - Birmingham Gastroenterology Associates, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Digestive Health Specialists of the Southeast, PA, Dothan, Alabama
  - Mayo Clinic, Phoenix, Arizona
  - The University of Arizona, Tucson, Arizona
  - Advanced Clinical Research Institute, LLC, Anaheim, California
  - Franco Felizarta, MD, Bakersfield, California
  - Southern California Liver Centers, Coronado, California
  - West Coast Clinical Trials, LLC, Costa Mesa, California
  - Scripps Clinic Medical Group, La Jolla, California
  - eStudySite, La Mesa, California
  - Long Beach VA Medical Center, Long Beach, California
  - Ruane Clinical Research Group, Los Angeles, California
  - National Research Institute, Los Angeles, California
  - Anthony Mills MD, Inc, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente, Los Angeles, California
  - Veterans Administration Wadsworth Medical Center, Los Angeles, California
  - eStudySite, Oceanside, California
  - Stanford University, Palo Alto, California
  - Huntington Medical Research Institutes, Pasadena, California
  - Inland Empire Liver Foundation, Rialto, California
  - University of California Davis Medical Center, Sacramento, California
  - UC Davis Medical Center, Sacramento, California
  - University of California at San Diego, San Diego, California
  - Research and Education, Inc., San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Kaiser Permanente, San Diego, California
  - University of California San Diego, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Quest Clinical Research, San Francisco, California
  - Kaiser Permanente Center, San Francisco, California
  - Silicon Valley Research Institute, San Jose, California
  - Los Angeles BioMedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Hospital, Aurora, Colorado
  - South Denver Gastroenterology, Englewood, Colorado
  - Gastroenterology Center of Connecticut, Hamden, Connecticut
  - Yale University, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Whitman-Walker Health, Washington D.C., District of Columbia
  - Capital Medical Associates, P.C., Washington D.C., District of Columbia
  - Bach and Godofsky Infectious Diseases, Bradenton, Florida
  - University of Miami - Dept of Neurology, Coral Gables, Florida
  - University of Florida Hepatology Research at CTRB, Gainesville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Saint Joseph's Hospital, Tampa, Florida
  - Tampa General Hospital, Tampa, Florida
  - South Florida Center of Gastroenterology, P.A., Wellington, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Atlanta Medical Center, Atlanta, Georgia
  - Dekalb Gastroenterology Associates, LLC, Decatur, Georgia
  - Infectious Disease Specialists of Atlanta, PC, Decatur, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - The Queen's Medical Center-Liver Center, Honolulu, Hawaii
  - Ruth M. Rothstein CORE Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Delta Research Partners, LLC, Bastrop, Louisiana
  - Medical Development Centers, LLC, Baton Rouge, Louisiana
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Digestive Disease Associates, PA, Baltimore, Maryland
  - University of Maryland, College Park, Maryland
  - Johns Hopkins University, Lutherville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Community Research Initiative of New England, Boston, Massachusetts
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Partners in Internal Medicine, PC, Worcester, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Minnesota Gastroenterology, Saint Paul, Minnesota
  - Digestive Health Specialists, Tupelo, Mississippi
  - Kansas City Research Institute, LLC, Kansas City, Missouri
  - The Kansas City Free Health Clinic, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Saint Louis University, St Louis, Missouri
  - Comprehensive Clinical Research, Berlin, New Jersey
  - ID Care, Inc., Hillsborough, New Jersey
  - Atlantic Research Affiliates, LLC, Morristown, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - The Gastroenterology Group of South Jersey, Vineland, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Southwest C.A.R.E. Center, Santa Fe, New Mexico
  - Binghamton Gastroenterology Associates, PC, Binghamton, New York
  - Northwell Health, Manhasset, New York
  - Concorde Medical Group PLLC, New York, New York
  - Weill Cornell Medical College of Cornell Univeristy, New York, New York
  - St. Luke's Roosevelt Hospital, New York, New York
  - Columbia Presbyterian Hospital, Columbia University, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester, Rochester, New York
  - Bronx Veteran's Affairs Medical Center, The Bronx, New York
  - Westchester Digestive Disease Group, Yonkers, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Carolinas Center for Liver Disease, Statesville, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Options Health Research LLC, Tulsa, Oklahoma
  - Schleinitz Research and Gastroenterology LLC, Medford, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Lehigh Valley Health Network, Network Office of Research and Innovation, Allentown, Pennsylvania
  - Regional Gastroenterology Associates of Lancaster, Ltd., Lancaster, Pennsylvania
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - UPMC Center For Liver Diseases, Pittsburgh, Pennsylvania
  - Veterans Affairs Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - Gastro One, Germantown, Tennessee
  - The Frist Clinic, Nashville, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Quality Medical Research, PLLC, Nashville, Tennessee
  - The North Texas Clinical Research Institute, Arlington, Texas
  - Central Texas Clinical Research, LLC, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor Endocrine Center, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Methodist Dallas Medical Center, Dallas, Texas
  - Southwest Infectious Disease Clinical Research, Inc, Dallas, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Kelsey Research Foundation, Houston, Texas
  - Research Specialists of Texas, Houston, Texas
  - St. Luke's Health Baylor College of Medicine Medical Center, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - CHI Health Reseach Center, Houston, Texas
  - Gastroenterology Consultants PLC, Live Oak, Texas
  - The Texas Liver Institute, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - PRA Health Sciences, Salt Lake City, Utah
  - Metropolitan Research, Annandale, Virginia
  - Inova Fairfax Hospital Center for Liver Diseases, Falls Church, Virginia
  - Liver Institute of Virginia, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Australia (24):
  - Canberra Specialist Centre, Canberra, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - East Sydney Doctors, Darlinghurst, New South Wales
  - Holdsworth House Medical Practice, Darlinghurst, New South Wales
  - St Vincent's Public Hospital Sydney, Darlinghurst, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders University, Bedford Park, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Footscray Hospital, Footscray, Victoria
  - Austin Health, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Greenslopes Private Hospital, Greenslopes
  - Royal Brisbane & Women's Hospital, Herston
  - Sir Charles Gairdner Hospital, Nedlands
  - Royal Perth Hospital, Perth
  - Princess Alexandra Hospital, Woolloongabba
- Austria (3):
  - Medizinische Universität Graz, Graz, Styria
  - Medizinische Universität Wien, Vienna, Vienna
  - Wilhelminenspital der Stadt Wien, Vienna, Vienna
- Belgium (4):
  - Ziekenhuis Netwerk Antwerpen Campus Stuivenberg, Antwerp
  - Cliniques Universitaires Saint Luc, Brussels
  - Université Libre de Bruxelles Hôpital Erasme, Brussels
  - AZ Groeninge Kortrijk, Kortrijk
- Canada (12):
  - University of Calgary Liver Unit, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Liver and Intestinal Research Center, Vancouver, British Columbia
  - GIRI GI Research Institute, Vancouver, British Columbia
  - Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Vancouver Infectious Disease Research and Care Centre, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Ottawa General Hospital, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Centre Hospitalier de L'Universite de Montreal (CHUM), Montreal, Quebec
- Czechia (3):
  - Slezska nemocnice v Opave, Infekcni oddeleni, Opava
  - Klin med, s.r.o., Prague
  - Remedis, s.r.o., Prague
- Estonia (2):
  - West Tallinn Central Hospital, Talinn
  - Tartu University Hospital, Tartu
- France (23):
  - Centre Hospitalier Universitaire de Grenoble, Cedex 9, Auvergne-Rhône-Alpes
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand, Auvergne
  - Hôpital Claude Huriez- Service d'Hépato-Gastroentérologie, Lille, Hauts-de-France
  - Hopitaux De Brabois, Vandœuvre-lès-Nancy, Limousin, Lorraine
  - Centre Hospitalier Universitaire (CHU) De Limoges - Hopital Dupuytren, Limoges, Limousin
  - CIC Hopital Purpan, Toulouse, Midi-pyrenees
  - Hôpital-Saint Joseph, Service D'Hépato-Gastroentérologie, Marseille, Provence-Alpes-Côte d'Azur Region
  - Hôpital de I´Archet 2, Nice, Provence-Alpes-Côte d'Azur Region
  - Hopital Beaujon, Clichy
  - Hopital Saint-Eloi, Montpellier
  - CHU de Nice - Hôpital l'Archet, Nice
  - Hôpital Saint Louis, Paris
  - Hôpital la Pitié Salpêtrière, Paris
  - Hôpital Cochin, Paris
  - Centre Hospitalier Universitaire Bordeaux Hôpital Haut-Lévêque, Pessac
  - Hopital Pontchaillou, Rennes
  - C.H.U. Strasbourg, Strasbourg
  - Hôpital Henri Mondor, Créteil, Île-de-France Region
  - Hôpital Saint-Antoine, Paris, Île-de-France Region
  - CHU Pitié-Salpêtrière, Paris, Île-de-France Region
  - Hôpital Bichat-Claude Bernard, Paris, Île-de-France Region
  - Hôpital Tenon, Paris, Île-de-France Region
  - Hôpital Paul Brousse, Villejuif, Île-de-France Region
- Germany (24):
  - Albert-Ludwigs-Universität, Freiburg im Breisgau, Baden-Wurttemberg
  - PraxisZentrum für Gastroenterologie und Endokrinologie, Freiburg im Breisgau, Baden-Wurttemberg
  - Medizinische Universitätsklinik IV (Krehl Klinik) Abt. Gastroenterologie und Infektionskrankhen, Heidelberg, Baden-Wurttemberg
  - Medizinische Klinik und Poliklinik III, München, Bavaria
  - Infektiologikum Frankfurt, Frankfurt am Main, Hesse
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Klinikum der Universität zu Köln, Cologne, North Rhine-Westphalia
  - Medizinisches Versorgungszentrum, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Gastroenterologische Gemeinschaftspraxis, Herne, North Rhine-Westphalia
  - Centrum für Interdisziplinäre Medizin, Münster, North Rhine-Westphalia
  - Leber- and Studienzentrum am Checkpoint, Berlin
  - EPIMED GmbH, Berlin
  - Charité Universitätsmedizin Berlin, Berlin
  - Zentrum für Infektiologie Berlin Prenzlauer Berg GmbH, Berlin
  - Universitäts Bonn, Bonn
  - Universitätsklinikum Frankfurt, Frankfurt
  - Asklepios Klinik St. Georg, Hamburg
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Gastroenterologische Gemeinschaftspraxis Kiel Preetzer, Kiel
  - University of Leipzig, Leipzig
  - Mainz University, Mainz
- Italy (15):
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera di Bologna - Policlinico S. Orsola Malpighi, Bologna
  - Azienda Ospedaliera S. Orsola - Malpighi, Bologna
  - Ente Ospedaliero Ospedali Galliera di Genova, Genova
  - Ospedale San Raffaele-IRCCS, Centro San Luigi - San Raffaele Turro, Unità Operativa di Malattie Infettive, Milan
  - Azienda Ospedaliera - Polo Universitario Luigi Saco, Milan
  - Azienda Ospedaliera Ospedale Niguarda Ca' Granda, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Padova, U.O.C. Cardiologia, Padua
  - Azienda Ospedaliera-universitaria Policlinico P. Giaccone, Palermo
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Instituto Nationale Per Le Malattie Infettive "Lazzaro Spallanzani", Roma
  - Fondazione Policlinico Tor Vergata, Roma
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Netherlands (4):
  - Academisch Medisch Centrum, Amsterdam, North Holland
  - Leiden Universitair Medisch Centrum, Leiden, South Holland
  - Erasmus Medisch Centrum, Rotterdam, South Holland
  - Universitair Medisch Centrum Sint Radboud, Nijmegen
- New Zealand (7):
  - Auckland Clinical Studies Limited, Grafton, Auckland
  - Auckland City Hospital, Grafton, Auckland
  - Bay of Plenty Clinical School, Tauranga, Bay of Plenty
  - Wellington Hospital, Newtown, WGN
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Urosurgery, Hamilton
- Poland (6):
  - Centrum Badan Klinicznych, Wroclaw, Lower Silesian Voivodeship
  - SP ZOZ Wojewódzki Szpital Zakazny, Warsaw, Masovian Voivodeship
  - Wojewódzki Szpital Specjalistyczny im. Kazimierza Dluskiego w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Szpital Specjalistyczny w Chorzowie, Chorzów, Silesian Voivodeship
  - ID Clinic Arkadiusz Pisula, Mysłowice, Silesian Voivodeship
  - Spzoz Wojewodzki Specjalistyczny Szpital im. W. Bieganskiego W Lodzi, Lodz
- Puerto Rico (2):
  - Clinical Research Puerto Rico, San Juan, PR
  - Fundacion De Investigacion De Diego, San Juan
- Spain (10):
  - Hospital Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga, Malaga
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Nuestra Señora de Valme, Seville
  - Hospital General Universitario de Valencia, Valencia
- Sweden (4):
  - Sahlgrenska Universitetssjukhuset, Östra Sjukhus, Gothenburg
  - Skånes Universitetssjukhus i Lund, Lund
  - Skånes Universitetssjukhus,, Malmo
  - Karolinska University Hospital Huddinge, Stockholm
- United Kingdom (14):
  - University of Birmingham and Queen Elizabeth Hospital Birmingham, Birmingham, England
  - Bristol Royal Infirmary, Bristol, England
  - St George Hospital, London, England
  - Chelsea and Westminster Hospital NHS Foundation Trust, London, England
  - Guy's and Saint Thomas NHS Foundation Trust, London, England
  - Imperial College Healthcare NHS Trust, London, England
  - King's College Hospital, London, England
  - Royal Free London NHS Foundation Trust, London, England
  - North Manchester General Hospital, Manchester, England
  - Nottingham University Hospitals NHS Trust, Nottingham, England
  - John Radcliffe Hospital, Oxford, England
  - Derriford Hospital, Plymouth, England
  - Queen Alexandra Hospital, Portsmouth, England
  - Southampton University Hospitals NHS Trust, Southampton General Hospital, Southampton, England

REFERENCES:
- [Derived] Younossi ZM, Stepanova M, Racila A, Afendy A, Lawitz EJ, Schwabe C, Ruane PJ, Lalezari J, Reddy KR, Jacobson IM, Muir AJ, Gaggar A, Myers RP, Younossi I, Nader F. Long-term Benefits of Sustained Virologic Response for Patient-Reported Outcomes in Patients With Chronic Hepatitis C Virus Infection. Clin Gastroenterol Hepatol. 2020 Feb;18(2):468-476.e11. doi: 10.1016/j.cgh.2019.07.047. Epub 2019 Jul 31. PMID 31376493